CLINICAL TRIAL: NCT06857396
Title: Tracheal Exposure Without Tracheostomy Completion : a New Protocol for Airway Management in Trans-oral Robotic Oncologic Surgery
Brief Title: Tracheal Exposure Without Tracheostomy Completion in Trans-oral Robotic Oncologic Surgery
Acronym: TRACH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-004
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Upper Aerodigestive Tract Neoplasms
Keywords: Tracheostomy; Upper aerodigestive tract neoplasms; Robotic-assisted surgery; Unnecessary surgery; Surgery complications
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREPA-TRACH Patient cohort: Patients included in the PREPA TRACH surgery protocol
  Interventions: Procedure: PREPA-TRACH

INTERVENTIONS:
Procedure: PREPA-TRACH — Tracheal exposure without tracheostomy completion during trans-oral robotic oncologic surgery

SUMMARY:
Upper aerodigestive tract neoplasms surgery results in important trauma, including swelling (oedemas) that can lead to respiratory tract obstruction and death from suffocation. To prevent this, protective tracheostomy is performed, allowing patients to breathe through a cannula during the critical phase. Although tracheostomy is reassuring, it presents complications, including swallowing disorders, refeeding delay and pulmonary infections. It generates anxiety for patients and can prevent them from communicating, which can affect their psychological well-being during hospitalization.

In Sainte Musse Hospital, patients who undergo upper aerodigestive tract neoplasms surgery are continuously monitored in intensive care unit. For some "at risk" patients, tracheostomy preparation is performed during operation with tracheal exposure but no incision. If dyspnea occurs, reanimators can quickly access to trachea and proceed to tracheostomy completion. This method, called PREPA-TRACH, avoids unnecessary tracheostomies while minimizing risks for the patients who would need it. Study purpose is to assess the security and reliability of this PREPA-TRACH protocol.

DETAILED DESCRIPTION:
This retrospective descriptive monocentric study aims at producing a descriptive series of patients who underwent tracheal exposure in case of tracheostomy hoping to avoid them a complete tracheostomy. Its purpose is to demonstrate on one hand the reliability and security of this technique and on the other hand to define some imperative criteria of surgical indication for tracheostomy or no tracheostomy. The number of patients included corresponds to the eligible patients cohort of Hôpital Sainte Musse ENT surgery department over the 10 last years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* All patients managed for an upper airway and digestive tract carcinoma with trans-oral robotic surgery, with tracheal exposure performed during the surgical procedure without immediate tracheostomy completion.

Exclusion Criteria:

* Patients with immediate complete laryngectomy or complete pharyngolaryngectomy
* Patient opposition
* Patient under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed for an upper airway and digestive tract carcinoma with a trans-oral robotic surgery with tracheal exposure performed during the surgical procedure without immediate tracheotomy completion.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Tracheostomy completion rate | Up to 3 hours
  The number of post-operatory complete tracheostomies finally performed over the total number of patients included in the PREPA-TRACH protocol will be calculated.

SECONDARY OUTCOMES:
Overall survival rate | Up to 3 hours
  Number of patients included in the PREPA-TRACH protocol who died because of post-operatory asphyxia.
Hospital length of stay | Up to 3 weeks
  Average hospital length of stay will be calculated depending on whether tracheostomy was finally performed or not.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume ROUGIER, MD, Study Director — CHITS
Locations (1):
- ENT and oncologic surgery department, Sainte-Musse Hospital, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poissonnet V, Chabrillac E, Schultz P, Moriniere S, Gorphe P, Baujat B, Garrel R, Lasne-Cardon A, Villeneuve A, Chambon G, Fakhry N, Aubry K, Dufour X, Malard O, Mastronicola R, Vairel B, Gallet P, Ceruse P, Jegoux F, Ton Van J, De Bonnecaze G, Vergez S. Airway management during transoral robotic surgery for head and neck cancers: a French GETTEC group survey. Eur Arch Otorhinolaryngol. 2022 Jul;279(7):3619-3627. doi: 10.1007/s00405-021-07188-4. Epub 2022 Jan 23. PMID 35066651
- [Background] Mandal R, Duvvuri U, Ferris RL, Kaffenberger TM, Choby GW, Kim S. Analysis of post-transoral robotic-assisted surgery hemorrhage: Frequency, outcomes, and prevention. Head Neck. 2016 Apr;38 Suppl 1:E776-82. doi: 10.1002/hed.24101. Epub 2015 Jul 15. PMID 25916790